CLINICAL TRIAL: NCT06318273
Title: A Phase 1 First-in-Human Study Evaluating Safety, Pharmacokinetics, and Efficacy of ABBV-969 in Adult Subjects With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study to Assess Adverse Events, and How Intravenously (IV) Infused ABBV-969 Moves Through the Bodies of Adult Participants With Metastatic Castration-Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M24-742; 2024-516772-15-00 (Other: EU CT)
Record Dates: First submitted 2024-03-13; First posted 2024-03-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: Metastatic Castration-Resistant Prostate Cancer; mCRPC; ABBV-969

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part 1: ABBV-969 Dose Escalation (Experimental): Participants will receive escalating doses of ABBV-969.
  Interventions: Drug: ABBV-969
- Part 2 A: ABBV-969 Dose Expansion (Experimental): Participants will receive dose A of ABBV-969 from part 1.
  Interventions: Drug: ABBV-969
- Part 2 B: ABBV-969 Dose Expansion (Experimental): Participants will receive dose B of ABBV-969 from part 1.
  Interventions: Drug: ABBV-969

INTERVENTIONS:
Drug: ABBV-969 — Intravenous (IV) Infusion

SUMMARY:
Prostate cancer has the second highest incidence rate and is the fifth leading cause of cancer-related deaths among men worldwide. The purpose of this study is to assess safety, pharmacokinetics, and efficacy of ABBV-969 as a monotherapy.

ABBV-969 is an investigational drug being developed for the treatment of metastatic castration-resistant prostate cancer (mCRPC). There are parts to this study. Participants will receive ABBV-969 as a single agent at different doses. Approximately 140 adult participants will be enrolled in the study across sites worldwide.

In part 1 (dose escalation), ABBV-969 will be intravenously infused in escalating doses as a monotherapy. In part 2, multiple doses will be selected from Part 1 and mCRPC participants will be assigned to one of these doses in a randomized fashion to determine the recommended Phase 2 dose. The estimated duration of the study is up to 3 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic and may require frequent medical assessments, blood tests, and scans.

ELIGIBILITY:
Inclusion Criteria:

* Histological, pathological, and/or cytological confirmation of adenocarcinoma of the prostate.
* Estimated life expectancy > 6 months.
* Must have progressed on prior novel hormonal agents (NHAs) (e.g., abiraterone acetate and/or enzalutamide) for the treatment of metastatic prostate cancer and/or castration-resistant prostate cancer (CRPC). Determination of progression is done per local investigator according to Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1 and/or Prostate Cancer Working Group 3 (PCWG3).
* Serum testosterone levels <= 50 ng/dL (<= 1.73 nmol/L) within the screening period and prior to the first dose of the study drug.
* Must have received at least one NHA (e.g., enzalutamide and/or abiraterone). Additionally, participants must have received at least one taxane for prostate cancer (or have refused, or are intolerant to, or unable to get access to taxanes).
* Must have >= 1 metastatic lesion that is present on baseline computed tomography (CT), magnetic resonance imaging (MRI), or bone scan imaging obtained <= 28 days prior to beginning study therapy.
* Serum prostate specific antigen (PSA) level >= 1.0 ng/mL.
* Availability of representative baseline tumor tissue (most recent archived tumor tissue after any novel hormonal agent (NHA) and/or any Prostate-Specific Membrane Antigen (PSMA) targeted therapy or fresh biopsy collected during screening phase) suitable for immunohistochemistry (IHC) testing. This requirement may be waived at the discretion of the AbbVie Medical Monitor if collecting a biopsy at screening would place the subject at risk of harm or would require a technically complicated procedure based on tumor location as assessed by the investigator.
* Laboratory values meeting the criteria laid out in the protocol.
* QT interval corrected for heart rate (QTc) <= 470 msec (using Fridericia's correction), no >= Grade 3 arrythmia, and no other clinically significant cardiac abnormalities.

Exclusion Criteria:

* Unresolved Grade 2 or higher toxicities related to previous anticancer therapy except alopecia.
* History of other active malignancy, as laid out in the protocol.
* History of interstitial lung disease (ILD) or pneumonitis that required treatment with systemic steroids, nor any evidence of active ILD or pneumonitis on screening chest CT scan.
* History of or active idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis.
* History of or active clinically significant, intercurrent lung-specific illnesses including, but not limited to those listed in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Up to 3 Years
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.
Percentage of Participants Achieving Prostate Specific Antigen (PSA) response | Up to 3 Years
  PSA response is defined as >= 50% PSA decrease from baseline.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of ABBV-969 | Up to 3 Years
  Cmax is defined as the maximum observed plasma/serum concentration of ABBV-969.
Time to Maximum Observed Concentration (Tmax) of ABBV-969 | Up to 3 Years
  Tmax is defined as the time to maximum observed concentration of ABBV-969.
Terminal Phase Elimination Half-Life (t1/2) of ABBV-969 | Up to 3 Years
  Terminal phase elimination half-life of ABBV-969.
Area Under the Plasma/Serum Concentration Versus Time Curve (AUC) of ABBV-969 | Up to 3 Years
  Area under the plasma/serum concentration versus time curve (AUC) of ABBV-969.
Antidrug Antibody (ADA) | Up to 3 Years
  Incidence and concentration of anti-drug antibodies.
Neutralizing Antibodies (nAbs) | Up to 3 Years
  Incidence and concentration of neutralizing antibodies.
Recommended Phase 2 Dose (RP2D) of ABBV-969 (Dose-Escalation Phase) | Up to 2 Years
  The RP2D of ABBV-969 will be determined during the dose-escalation phase of the study. RP2D will be determined using available safety and pharmacokinetics and pharmacodynamics data.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (26):
- United States (9):
  - City of Hope /ID# 262059, Duarte, California
  - Univ California, San Francisco /ID# 261715, San Francisco, California
  - Yale University School of Medicine /ID# 262234, New Haven, Connecticut
  - AdventHealth Orlando /ID# 261686, Orlando, Florida
  - University of Chicago Medical Center /ID# 261605, Chicago, Illinois
  - START Midwest /ID# 264295, Grand Rapids, Michigan
  - Carolina BioOncology Institute /ID# 261602, Huntersville, North Carolina
  - Lifespan Cancer Institute at Rhode Island Hospital /ID# 261687, Providence, Rhode Island
  - NEXT Oncology /ID# 261601, San Antonio, Texas
- Australia (3):
  - Chris O'Brien Lifehouse /ID# 261731, Camperdown, New South Wales
  - Ballarat Base Hospital /ID# 264294, Ballarat, Victoria
  - St Vincent's Hospital /ID# 264293, Fitzroy, Victoria
- Canada (2):
  - Centre Hospitalier de l'Université de Montréal (CHUM) /ID# 270890, Montreal, Quebec
  - McGill University Health Centre - Glen Site. /ID# 271275, Montreal, Quebec
- France (3):
  - Centre Oscar Lambret /ID# 270602, Lille, Nord
  - Centre Leon Berard /ID# 270605, Lyon, Rhone
  - Institut Gustave Roussy /ID# 270603, Villejuif, Île-de-France Region
- Israel (3):
  - The Chaim Sheba Medical Center /ID# 261772, Ramat Gan, Tel Aviv
  - Rambam Health Care Campus- Haifa /ID# 261770, Haifa
  - Hadassah Medical Center-Hebrew University /ID# 261771, Jerusalem
- Japan (3):
  - National Cancer Center Hospital East /ID# 261606, Kashiwa-shi, Chiba
  - Kyoto University Hospital /ID# 261861, Kyoto, Kyoto
  - National Cancer Center Hospital /ID# 261698, Chuo-ku, Tokyo
- Spain (3):
  - Hospital Universitario Vall de Hebron /ID# 270889, Barcelona
  - Hospital Universitario HM Sanchinarro /ID# 271345, Madrid
  - Hospital Universitario Virgen del Rocio /ID# 270617, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-742